CLINICAL TRIAL: NCT02154321
Title: EEG and ADHD Study
Brief Title: Electroencephalogram and Attention Deficit Hyperactivity Disorder Study
Status: Withdrawn | Type: Observational
Why Stopped: Funding and resource restrictions.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Chandra Sekhar Sripada, Chandra Sekhar Sripada, MD, PhD, University of Michigan
Other Study IDs: HUM00081947
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Attention Deficit Hyperactivity Disorder; Healthy Controls
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Attention Deficit Hyperactivity Disorder: This study aims to recruit 100 adult participants: 50 of which are adults diagnosed with Attention Deficit Hyperactivity Disorder and 50 healthy controls. All participants will perform a total of two tasks while connected to electroencephalogram (EEG) sensors; the first task is a resting state task and after that a cognitive challenge task (attention control). Study activity is performed in a single visit which lasts two hours. Participants will also be asked to complete some behavioral questionnaires.
  Interventions: Device: Electroencephalogram (EEG)
- Healthy Control: This study aims to recruit 100 adult participants: 50 of which are adults diagnosed with Attention Deficit Hyperactivity Disorder and 50 healthy controls. All participants will perform a total of two tasks while connected to electroencephalogram (EEG) sensors; the first task is a resting state task and after that a cognitive challenge task (attention control). Study activity is performed in a single visit which lasts two hours. Participants will also be asked to complete some behavioral questionnaires.
  Interventions: Device: Electroencephalogram (EEG)

INTERVENTIONS:
Device: Electroencephalogram (EEG) — The electroencephalogram assesses brain electrical activity through surface recording disks (electrodes) which are placed near the participants' head using a custom designed Lycra cap. The electrodes transmit the signals which are then amplified and stored on a computer. The procedure is entirely non-invasive. Once an accurate signal is assured, the signal derived from the electrode cap is then amplified, transmitted to a computer, and stored for later analysis. Each participant will undergo the electroencephalogram (EEG) procedure only once for the duration of 30-45 minutes.
  Other Names: ActiveTwo EEG System; Manufacturer: BioSemi; Supplier: Cortech Solutions; BEU Number: 409917

SUMMARY:
The purpose of this research is to assess and determine brain oscillations or "brain signatures" of adult participants with Attention Deficit Hyperactivity Disorder (ADHD) relative to adult participants without ADHD using the technique electroencephalogram (EEG). Electroencephalogram is entirely non-invasive way of tracking brain activity.The main goal of this study is to establish biological factors for determining the diagnosis of Attention Deficit Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria for all:

* Right-handedness

Inclusion Criteria for Attention Deficit Hyperactivity Disorder (ADHD) group:

* Currently unmedicated adults with ADHD. To be given a full diagnosis of adult ADHD, the participant must have full Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-R) criteria: (1) described a chronic course of ADHD symptomatology from childhood to adulthood, and (2) endorsed a moderate or sever level of impairment attributed to the ADHD symptoms.

Exclusion Criteria for all:

* Currently taking psychoative medications
* Any clinically significant neurological problem (e.g., tics, seizures, serious head injury)
* Alcohol or substance abuse (current or in the past 2 years)
* Any current Axis I psychiatric diagnosis (other than ADHD) as verified by clinical interview

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 adult participants will be recruited for this study: 50 adults diagnosed with Attention Deficit Hyperactivity Disorder and 50 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Brain Wave Measurements | Two years
  Measurement of electroencephalogram amplitude and coherence in alpha, gamma, and theta brain wave bands.

SECONDARY OUTCOMES:
Default Network Signatures | two years
  Measurement of the brain's default network consisting of interconnected midline and lateral parietal regions involved in internally directed mentation.

OTHER OUTCOMES:
Comparison of dependent measurements between Attention Deficit Hyperactivity Disorder and healthy controls | two years
  Comparison of dependent measures (i.e., computer tasks performed during electroencephalogram [EEG]: the Resting task and the Attention Control Task) between Attention Deficit Hyperactivity Disorder and healthy controls with independent sample t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra S Sripada, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- Rachel Upjohn Building, Ann Arbor, Michigan, United States